CLINICAL TRIAL: NCT02971020
Title: Proposal for Collection of Patient Data to Aid in Design of an Observational Study (i.e. Preparatory to Research) Evaluating Risk of Cognitive Impairment After Surgical and Transcatheter Valve Replacement.
Brief Title: Evaluating the Risk of Cognitive Impairment After Surgical and Transcatheter Aortic Valve Replacement
Acronym: CAVIAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minnesota Veterans Medical Research and Education Foundation (Other)
Collaborators: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Santiago Garcia, MD, Minnesota Veterans Medical Research and Education Foundation
Organization: Center for Veterans Research and Education (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 4588-A
Record Dates: First submitted 2016-09-12; First posted 2016-11-22 (Estimated); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Cardiovascular Disease; Aortic Valve Stenosis; Cognitive Assessments; Valve Surgery; Transcatheter Valve Replacement; Surgical Valve Replacement
MeSH Terms: conditions — Cardiovascular Diseases; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgical Aortic Valve Replacement (Other): Montreal Cognitive Assessment (MoCA); Trail Making Test Part A; Trail Making Test Part B; Phonemic Fluency (letter fluency) and Semantic Fluency (category).
  Interventions: Other: Observational/Cognitive Assessment
- Transcatheter Aortic Valve Replacement (Other): Montreal Cognitive Assessment (MoCA); Trail Making Test Part A; Trail Making Test Part B; Phonemic Fluency (letter fluency) and Semantic Fluency (category).
  Interventions: Other: Observational/Cognitive Assessment

INTERVENTIONS:
Other: Observational/Cognitive Assessment — Montreal Cognitive Assessment (MoCA); Trail Making Test Part A; Trail Making Test Part B; Phonemic Fluency (letter fluency) and Semantic Fluency (category).

SUMMARY:
The investigators are conducting a pilot study to compare cognitive outcomes among Veterans with severe aortic valve stenosis who are scheduled to undergo either aortic valve replacement.

DETAILED DESCRIPTION:
The investigators are conducting a pilot study to compare cognitive outcomes in up to 60 Veterans with severe aortic valve stenosis who are scheduled to undergo either transcatheter aortic valve replacement (TAVR) or surgical aortic valve replacement (SAVR) at the Minneapolis VA Health Care System. Participants will be administered a short battery of cognitive tests before and three months after TAVR or SAVR over/up to a two year study period.

ELIGIBILITY:
Inclusion Criteria:

* Severe aortic stenosis (AVA: 1 cm2 and/or mean gradient =or > 40 mmHg and/or peak velocity > 4 m/s)
* Scheduled to undergo either surgical or transcatheter aortic valve replacement at the Minneapolis VA Health Care System

Exclusion Criteria:

* Severe cognitive impairment at baseline (i.e. unable to understand or follow-up study procedures)
* Unable or unwilling to provide informed consent

Max Age: 104 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-11-12 (Actual); Study Completion 2018-03-21 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment | Three Months
  Estimate the means and standard deviations of changes in selected cognitive measures between baseline (pre-TAVR or pre-SAVR) and 3 months post-TAVR or post-SAVR, identify baseline correlates of those changes, and characterize baseline cognitive function and cognitive history of patients who undergo TAVR or SAVR.
Trail Making | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Garcia, MD, Principal Investigator — Minneapolis Veterans Affairs Medical Center; Howard Fink, MD, Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No